CLINICAL TRIAL: NCT00689780
Title: A Phase I, Multi-Centre, Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of AZD1940, Including an Interaction Study, After Administration of Oral Multiple Ascending Doses in Adult Subjects With Chronic Low Back Pain
Brief Title: Study to Investigate the Safety, Tolerability and Pharmacokinetics of AZD1940
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, AstraZeneca R&D Södertälje
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3120C00003
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Low Back Pain
Keywords: Pain; safety; chronic low back pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — N-(2-tert-butyl-1-((4,4-difluorocyclohexyl)methyl)-1H-benzo(d)imidazol-5-yl)ethanesulfonamide; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD1940 + Placebo
  Interventions: Drug: AZD1940
- 2 (Other)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: AZD1940 — Oral solution Multiple ascending dose given orally once daily at day 1-12
  Arms: 1
Drug: Midazolam — Oral solution given orally once daily on day -1 and day 14
  Arms: 2

SUMMARY:
A Phase I, Multi-Centre, Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of AZD1940, Including an Interaction Study, After Administration of Oral Multiple Ascending Doses in Adult Subjects with Chronic Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Chronic Low Back Pain according to Quebec Task force Class 1-3 and an average pain intensity score of 3-9 on NRS(0-10) during the past week.
* Clinical normal physical findings, including blood pressure, pulse rate > 45bpm, ECG (with normal QTcF interval <450msec and without any additional risk factors for Torsades de Pointes) and laboratory assessments, as judged by investigator
* Body Mass Index (BMI) ≥18 to ≤32 kg/m2 inclusive and body weight ≥50 to ≤100 kg

Exclusion Criteria:

* History of somatic disease/condition which may interfere with the objectives of the study, with the exception of Chronic Low Back Pain
* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder
* Clinically significant illness with the exception of Chronic Low Back Pain

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs) occurring during the study, blood pressure (supine and standing), pulse rate, respiratory rate, body temperature, laboratory variables and ECG | Vital signs, laboratory variables and adverse event each day throughout the study Paper printout ECG and/or digital ECG throughout the study

SECONDARY OUTCOMES:
Assessment of psychometric rating scales ( VAMS, CDR test battery, DEQ, ARCI and Bond-Lader) | Psychometric tests and VAMS (Visual Analogue Mood Scale) throughout the study
To investigate the PK profile (including dose proportionality) of AZD1940 by assessment of plasma concentrations | Bloodsampling Day 1,6, 10 and 15
Plasma levels of midazolam and 4ß hydroxycholesterol and 6β hydroxycortisol:cortisol urine excretion ratio as markers | Bloodsampling at day -1, 14

CONTACTS AND LOCATIONS:
Overall Officials: Janet Post, Study Chair — AstraZeneca R&D SödertäljeSE; Wolfgang Kühn, Principal Investigator — Quintiles AB Phase 1 Services Strandbodgatan Uppsala, Sweden+
Locations (3):
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Luleå
  - Research Site, Upssala